CLINICAL TRIAL: NCT07171502
Title: AI-Assisted Ultrasound-Guided Nerve Block: Model Development and Performance Assessment
Acronym: AI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Tao Xu, principal, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AI-Sacral Plexus
Record Dates: First submitted 2025-09-08; First posted 2025-09-12 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-09

CONDITIONS: AI (Artificial Intelligence); Ultrasound-Guided Nerve Blocks

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI Annotation (Experimental)
  Interventions: Device: AI Annotation
- Manual Annotation (Placebo Comparator)
  Interventions: Other: manual annotation

INTERVENTIONS:
Device: AI Annotation — Use the AI model to assist in annotating the target images.
  Arms: AI Annotation
Other: manual annotation — Use the manual to annotate the target images.
  Arms: Manual Annotation

SUMMARY:
This study intends to have experts with over 10 years of experience in ultrasound-guided regional anesthesia acquire 1,000 target images. These images will be annotated by both an AI model and human experts, and the model's annotations will be evaluated by a panel of 10 specialists. The primary outcome is the accuracy of identifying the target anatomical structures in the annotated images. Secondary outcomes include the number of true positive, false positive, true negative, and false negative structures, the time required for annotation, and the potential application of the AI model in assisting the performance of ultrasound-guided regional blocks.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years
* BMI between 19-23 kg·m-²
* ASA physical status classification I-II
* Normal orientation and able to cooperate with physical examination.

Exclusion Criteria:

* Patient refusal
* Infection, trauma, skin defect, deformity, or other abnormalities at the intended nerve block site
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2025-09-30 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
The accuracy of identifying the target anatomical structures in the annotated images. | From enrollment to the end of treatment at 4 months

SECONDARY OUTCOMES:
The number of true positive (TP) structures | From enrollment to the end of treatment at 4 months
The number of false positive (FP) structures | From enrollment to the end of treatment at 4 months
The number of true negative (TN) structures | From enrollment to the end of treatment at 4 months
The number of false negative (FN) structures | From enrollment to the end of treatment at 4 months
The annotation time (time from the start to the end of annotation) | From enrollment to the end of treatment at 4 months
An evaluation of the AI model if applied to assist in performing ultrasound-guided regional blocks: a) its impact on block failure rate (increase, no effect, decrease); b) its impact on the incidence of adverse events (increase, no effect, decrease) | From enrollment to the end of treatment at 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital Affiliated with Shanghai Jiao Tong University School of Medicine, Shanghai, China